CLINICAL TRIAL: NCT03895892
Title: The Effect of Exogenous Ketone Supplementation on 20 km Time Trial and Wingate Performance in Recreationally Active Individuals
Brief Title: Exogenous Ketone Supplementation and Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113474
Record Dates: First submitted 2019-02-13; First posted 2019-03-29 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Ketonemia; Ketosis
MeSH Terms: conditions — Ketosis | interventions — Ketones; Caffeine

STUDY DESIGN:
Intervention Model Description: This will be a double blind repeated measures cross over study. There will be three treatments involved: Caffeinated ketone supplements, non-caffeinated ketone supplement and water-placebo. Participants will complete the protocol three times and the treatment order will be systematically rotated to avoid any order effect. Design of the study is composed of two performance tests 30 minutes following supplementation. All participants will arrive in a fed state to the laboratory. the corresponding treatment will be provided and 30 minutes later, they will perform a 20 km time trial. 10 minutes after the time trial, participants will perform a 30 second all-out Wingate test.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded as an individual not involved in the project will assemble and distribute the treatment (drinks) according to a coding system that is kept confidential until the study is completed. Participants will complete the protocol three times and the treatment order will be systematically rotated to avoid any order effect. taste and texture of treatments will be matched and will be distribute in opaque bottles to keep participant blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Water Placebo (Placebo Comparator): Placebo flavored drink similar to treatments but with no energy will be ingested before completing a 20km Time trial and a 30 second all-out Wingate test
  Interventions: Behavioral: 20 km time trial; Behavioral: Wingate test; Dietary Supplement: Water Placebo
- Experimental 1 (Experimental): Ketone salts supplement mixed in water will be ingested before completing a 20km Time trial and a 30 second all-out Wingate test
  Interventions: Behavioral: 20 km time trial; Behavioral: Wingate test; Dietary Supplement: Ketone
- Experimental 2 (Experimental): Ketone salts/caffeine supplement mixed in water will be ingested before completing a 20km Time trial and a 30 second all-out Wingate test
  Interventions: Behavioral: 20 km time trial; Behavioral: Wingate test; Dietary Supplement: Ketone/Caffeine

INTERVENTIONS:
Behavioral: 20 km time trial — 20 km time trial cycling test will be conducted to measure the effect of different drinks on time
Behavioral: Wingate test — 30 second all-out effort on a bike will be conducted to measure the effect of different drinks on peak power output
Dietary Supplement: Ketone/Caffeine — Dietary supplement containing ketone salts and caffeine
  Arms: Experimental 2
Dietary Supplement: Ketone — Dietary supplement containing only ketone salts
  Arms: Experimental 1
Dietary Supplement: Water Placebo — Dietary supplement containing only water
  Arms: Water Placebo

SUMMARY:
20 healthy recreationally active men and woman aged 18-35 will participate in the study. There will be three treatments involved: Caffeinated ketone supplements, non-caffeinated ketone supplement and water-placebo. Participants will complete the protocol three times and the treatment order will be systematically rotated to avoid any order effect. The three main trials will be separated by at least 1 week. After providing the corresponding treatment, participants will be given 30 minutes and after, they will perform a standardized 10-minute warm-up, followed by the 20 km time trial and a 30-second all-out Wingate test.

DETAILED DESCRIPTION:
Some researchers support that a state of ketosis, reached through the use of ketogenic diet, has the potential to improve athletic. To attain such state, individuals must restrict carbohydrate intake to a maximum of 50g/ day or 10% while keeping protein intake moderate. One of the biggest challenges to achieve and maintain ketosis is complying with the diet due to its restrictive nature. Consequently, manufacturers have developed supplements that can induce a state of ketosis acutely (~1 hour). Unfortunately, there is very little evidence supporting the use of these supplements to enhance athletic performance. Hyperketonemia (blood ketone concentration > 0.2 Mm) seems to elevate the rate of utilization of ketone bodies. These changes in substrate utilization may allow athletes to preserve, something that would be advantageous for exercise performance. Ketone salts have been shown to elevate the concentration of ketones in blood and as such they may allow the body benefit from the apparent sparing of carbohydrates. Manufacturers now provide ketones salts combined with other ingredients such as caffeine. However it is unknown whether or not the addition of these ingredients has any positive or negative effect on athletic performance. Caffeine alone has been shown to improve athletic performance in several studies. Therefore, the purpose of this study is to compare the effectiveness of a caffeine free ketone salt supplement vs a caffeinated ketone salt supplement and their effects on a 20km time trial and a 30 second all-out Wingate test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female recreationally active individuals
* aged 15-35 years
* non regular caffeine users.

Exclusion Criteria:

* Smoker
* Taking part in other research
* Sedentary
* For women, if they are pregnant or become pregnant during the study
* Injury limiting exercise ability.
* Have symptoms or take medication for respiratory disease
* Have symptoms or take medication for cardiovascular disease
* Have symptoms or take mediation for neuromuscular disease
* Use heart rate or blood pressure medications
* Use any medications with side effects of dizziness, lack of motor control, or slowed reaction time

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
20 km time trial | 40 minutes
  participants will ride for 20 km on a stationary bike and time to complete distance will be measured.
Wingate test | 30 seconds
  participants will perform a ver short all-out effort on a stationary bike. peak power output and fatigue index will be measured.

SECONDARY OUTCOMES:
Blood Ketone | 1 hour
  blood ketones will be measured using ketone meter
Blood Lactate | 1 hour
  blood lactate will be measured using lactate meter
Rates of perceived exertion (RPE) | 1 hour
  RPE will be measured using Borg's scale (1= low - 10= high).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No